CLINICAL TRIAL: NCT00533650
Title: Proof of Concept (Bone Resorption/Bone Mineral Density) Study (0429-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0429-005; 2007_620
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-05

CONDITIONS: Post-Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — 3-(6-methoxypyridin-3-yl)-3-(2-oxo-3-(3-(5,6,7,8-tetrahydro(1,8)naphthyridin-2-yl)propyl)imidazolidin-1-yl)propionic acid

INTERVENTIONS:
Drug: MK0429

SUMMARY:
A study to asses the safety and efficacy of MK0429 in postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Person is a women with osteoporosis who is unwilling or unable to take other treatments for osteoporosis

Exclusion Criteria:

* Person has had a previous fracture
* Person has rheumatoid arthritis. Person has has certain types of cancer
* Person has donated blood or has been in another investigational study within the last 4 weeks

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2000-12; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC